CLINICAL TRIAL: NCT02559011
Title: Assessment of Arrhythmias in Patients Undergoing Transcatheter Aortic Valve Implantation Using a Small Insertable Cardiac Monitoring Device
Acronym: Reveal
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_09_21
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Aortic Valve Stenosis
Keywords: Arrhythmias, Cardiac; Transcatheter Aortic Valve implantation; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Patients who need a TAVI with symptomatic severe aortic valve stenosis

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has emerged as a valuable minimal-invasive treatment option in patients with symptomatic severe aortic valve (AV) stenosis at prohibitive or increased risk for conventional open-heart surgery. Recent randomized clinical trials reported a large treatment effect of TAVI over medical treatment among inoperable patients and similar or superior outcomes compared with surgical aortic valve replacement in high to intermediate risk patients. However, atrio-ventricular conduction disturbances and arrhythmias (in particular atrial fibrillation) before, during or after TAVI remain a matter of concern as they have important consequences.

The objective of this study is to investigate the incidence, nature and prognostic significance of AV-conduction disturbances and arrhythmias among patients with severe, symptomatic aortic stenosis undergoing TAVI before, during and after the procedure using a small implantable cardiac monitoring system (ICM; Medtronic REVEAL LinQTM).

One hundred patients will be enrolled in this study. Prior to TAVI (at least 4 weeks), at the time of preprocedural hemodynamic and anatomical assessment, the ICM will be inserted under the skin of the chest under local anesthesia. The device will be interrogated just prior to readmission for TAVI and thereafter at 1, 3, 6, and 12 months of follow-up. The incidence of symptomatic as well as silent brady- and tachyarrhythmias will be recorded, and its impact on medical and device treatment as well as clinical outcomes analyzed.

The present study will provide information about the actual incidence and impact of symptomatic and silent arrhythmias and AV-conduction disturbances among patients with severe, symptomatic aortic stenosis undergoing TAVI. Specifically, the study estimate the burden of arrhythmias before TAVI and to accurately determine the incidence of new onset atrial fibrillation and complete AV-block within 12 months after the procedure. Identifying patients at risk for AV- conduction abnormalities, atrial fibrillation (AF), and non-sustained or sustained ventricular arrhythmias may guide future preventive measures, medical treatment and improve patients outcomes after TAVI.

DETAILED DESCRIPTION:
Background

TAVI has emerged as a valuable minimal-invasive treatment option in patients with symptomatic severe aortic valve stenosis at prohibitive or increased risk for conventional open-heart surgery. AV conduction disturbances and arrhythmias before, during or after TAVI remain a matter of concern as they have consequences.

Prior to TAVI the ICM will be inserted under the skin of the chest under local anesthesia. The device will be interrogated just prior to readmission for TAVI and thereafter at 1, 3, 6, and 12 months of follow-up. The incidence of symptomatic as well as silent brady- and tachyarrhythmias will be recorded, and its impact on medical and device treatment as well as clinical outcomes analyzed.

All patients with severe, symptomatic aortic stenosis undergoing TAVI at the institution irrespective selected bioprosthesis will be included in the study. Final decision on eligibility will be made by the local Heart Team.

Objective

To investigate the incidence, nature and prognostic significance of AV-conduction disturbances and arrhythmias among patients with severe, symptomatic aortic stenosis undergoing TAVI before, during and after the procedure using a small implantable cardiac monitoring system (ICM; Medtronic REVEAL LinQTM). The primary endpoint of the study is to establish the incidence of new onset atrial fibrillation and complete AV-block within 12 months after TAVI.

Methods

One hundred patients with severe, symptomatic aortic stenosis undergoing TAVI will be enrolled in this prospective, observational study. Prior to TAVI (at least 4 weeks), at the time of preprocedural hemodynamic and anatomical assessment, the ICM will be inserted under the skin of the chest under local anesthesia. The device will be interrogated just prior to readmission for TAVI and thereafter at 1, 3, 6, and 12 months of follow-up. The incidence of symptomatic as well as silent brady- and tachyarrhythmias will be recorded, and its impact on medical and device treatment as well as clinical outcomes analyzed.

The study is observational: the patients will not be assigned to a specific intervention. Patients consenting will be monitored using a specific device that has been approved for market release. The objective of the study is to use the information obtained with this monitoring device to assess the incidence, nature and prognostic significance of atrioventricular conduction disturbances and arrhythmias among patients with severe, symptomatic aortic stenosis undergoing Transcatheter Aortic Valve Implantation before, during and after the procedure. The objective of the study is not to investigate the performance of the monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic valve stenosis undergoing TAVI

Exclusion Criteria

* Missing IC
* Pacemaker, internal cardioverter-defibrillator or cardiac resynchronization therapy (CRT) device at the time of screening
* Anatomic or clinical contraindications for TAVI or REVEAL insertion
* Patient currently participating in another study evaluating a new transcatheter valve prosthesis or a new drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with severe, symptomatic aortic valve stenosis undergoing TAVI at the institution irrespective selected bioprosthesis will be included in the study. Final decision on eligibility will be made by the local Heart Team.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with incidence of new onset atrial fibrillation and complete AVB within 12 months after TAVI | up to 12 months

SECONDARY OUTCOMES:
Number of patients with resolution of atrial Fibrillation | up to 12 months
Number of patients with resolution of Atrium Ventricular Block (AVB) after TAVI with permanent pacemaker (PPM) implantation | up to 12 months
Number of patients with cardiac death due to arrhythmias | up to 12 months
Number of patients with stroke | up to 12 months
Number of patients with presyncope and syncope | up to 12 months
Number of patients with pacemaker Implantation | up to 12 months
Number of patients with cardiovascular mortality | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Prof. Dr. med., Principal Investigator — Bern University Hospital, Dep. of Cardiology
Locations (1):
- Bern University Hospital, Dep. of Cardiology, Bern, Switzerland

REFERENCES:
- [Background] Mirabel M, Iung B, Baron G, Messika-Zeitoun D, Detaint D, Vanoverschelde JL, Butchart EG, Ravaud P, Vahanian A. What are the characteristics of patients with severe, symptomatic, mitral regurgitation who are denied surgery? Eur Heart J. 2007 Jun;28(11):1358-65. doi: 10.1093/eurheartj/ehm001. Epub 2007 Mar 9. PMID 17350971
- [Background] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Background] Friedman HS, Zaman Q, Haft JI, Melendez S. Assessment of atrioventricular conduction in aortic valve disease. Br Heart J. 1978 Aug;40(8):911-7. doi: 10.1136/hrt.40.8.911. PMID 687491
- [Background] Harris A, Davies M, Redwood D, Leatham A, Siddons H. Aetiology of chronic heart block. A clinico-pathological correlation in 65 cases. Br Heart J. 1969 Mar;31(2):206-18. doi: 10.1136/hrt.31.2.206. No abstract available. PMID 5775291
- [Background] Urena M, Hayek S, Cheema AN, Serra V, Amat-Santos IJ, Nombela-Franco L, Ribeiro HB, Allende R, Paradis JM, Dumont E, Thourani VH, Babaliaros V, Francisco Pascual J, Cortes C, Del Blanco BG, Philippon F, Lerakis S, Rodes-Cabau J. Arrhythmia burden in elderly patients with severe aortic stenosis as determined by continuous electrocardiographic recording: toward a better understanding of arrhythmic events after transcatheter aortic valve replacement. Circulation. 2015 Feb 3;131(5):469-77. doi: 10.1161/CIRCULATIONAHA.114.011929. Epub 2014 Dec 2. PMID 25466975
- [Background] Smith R, Grossman W, Johnson L, Segal H, Collins J, Dalen J. Arrhythmias following cardiac valve replacement. Circulation. 1972 May;45(5):1018-23. doi: 10.1161/01.cir.45.5.1018. No abstract available. PMID 5020795
- [Background] Matthews IG, Fazal IA, Bates MG, Turley AJ. In patients undergoing aortic valve replacement, what factors predict the requirement for permanent pacemaker implantation? Interact Cardiovasc Thorac Surg. 2011 Mar;12(3):475-9. doi: 10.1510/icvts.2010.254607. Epub 2010 Dec 7. PMID 21138915
- [Background] Moreno R, Dobarro D, Lopez de Sa E, Prieto M, Morales C, Calvo Orbe L, Moreno-Gomez I, Filgueiras D, Sanchez-Recalde A, Galeote G, Jimenez-Valero S, Lopez-Sendon JL. Cause of complete atrioventricular block after percutaneous aortic valve implantation: insights from a necropsy study. Circulation. 2009 Aug 4;120(5):e29-30. doi: 10.1161/CIRCULATIONAHA.109.849281. No abstract available. PMID 19652115
- [Background] Rubin JM, Avanzas P, del Valle R, Renilla A, Rios E, Calvo D, Lozano I, Anguera I, Diaz-Molina B, Cequier A, Moris de la Tassa C. Atrioventricular conduction disturbance characterization in transcatheter aortic valve implantation with the CoreValve prosthesis. Circ Cardiovasc Interv. 2011 Jun;4(3):280-6. doi: 10.1161/CIRCINTERVENTIONS.111.961649. Epub 2011 May 3. PMID 21540440
- [Background] Adams DH, Popma JJ, Reardon MJ. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 Sep 4;371(10):967-8. doi: 10.1056/NEJMc1408396. No abstract available. PMID 25184874
- [Background] van der Boon RM, Nuis RJ, Van Mieghem NM, Jordaens L, Rodes-Cabau J, van Domburg RT, Serruys PW, Anderson RH, de Jaegere PP. New conduction abnormalities after TAVI--frequency and causes. Nat Rev Cardiol. 2012 May 1;9(8):454-63. doi: 10.1038/nrcardio.2012.58. PMID 22547171
- [Background] Houthuizen P, Van Garsse LA, Poels TT, de Jaegere P, van der Boon RM, Swinkels BM, Ten Berg JM, van der Kley F, Schalij MJ, Baan J Jr, Cocchieri R, Brueren GR, van Straten AH, den Heijer P, Bentala M, van Ommen V, Kluin J, Stella PR, Prins MH, Maessen JG, Prinzen FW. Left bundle-branch block induced by transcatheter aortic valve implantation increases risk of death. Circulation. 2012 Aug 7;126(6):720-8. doi: 10.1161/CIRCULATIONAHA.112.101055. Epub 2012 Jul 12. PMID 22791865
- [Derived] Nozica N, Siontis GCM, Elchinova EG, Goulouti E, Asami M, Bartkowiak J, Baldinger S, Servatius H, Seiler J, Tanner H, Noti F, Haeberlin A, Branca M, Lanz J, Stortecky S, Pilgrim T, Windecker S, Reichlin T, Praz F, Roten L. Assessment of New Onset Arrhythmias After Transcatheter Aortic Valve Implantation Using an Implantable Cardiac Monitor. Front Cardiovasc Med. 2022 May 16;9:876546. doi: 10.3389/fcvm.2022.876546. eCollection 2022. PMID 35651903